CLINICAL TRIAL: NCT03836378
Title: Innovative Addition of Dehydrated Human Amnion-Chorion Membrane During Scaling and Root Planing
Brief Title: Addition of Dehydrated Human Amnion-Chorion Membrane During Scaling and Root Planing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 18-2447
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Diseases
Keywords: Non-surgical periodontal therapy; Outcomes; Clinical trial; Periodontitis; Academic setting
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: The participant will have half the mouth completed with scaling and root planing alone and half the mouth completed with scaling and root planing with the addition of membrane in deep probing depth sites.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A random allocation will be completed (flip of coin) which side will receive the membrane placement. The care provider (hygienist) will be aware of the membrane placement. The investigator and outcome assessor (periodontist) will not know which sites received the membrane placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Cleaning and Intervention (Experimental): One side of the participant's mouth will receive a deep cleaning in addition to the placement of a BioXclude™ membrane in the deep pocket sites. The participant will then be followed for 9 months with routine care.
  Interventions: Procedure: BioXclude™
- Deep Cleaning Only (No Intervention): One side of the participant's mouth will receive deep cleaning (scaling and root planning) only. The participant will then be followed for 9 months with routine care.

INTERVENTIONS:
Procedure: BioXclude™ — The addition of BioXclude™ dehydrated human amnion-chorion membrane into deep pockets with scaling and root planing.
  Arms: Deep Cleaning and Intervention

SUMMARY:
Hypothesis: There will be an additional reduction of pocket depth and gain of clinical attachment when dehydrated human amnion-chorion membrane (dHACM) is placed into the periodontal disease defect after mechanical scaling and root planing.

Specific Aim 1: to compare the clinical and radiographical outcome of using dehydrated human amnion-chorion membrane (dHACM) (commercially available as BioXclude®) with mechanical scaling and root planing.

DETAILED DESCRIPTION:
The study product BioXclude™ is a commercially available Amnion-Chorion allograft membrane. BioXclude™ does not meet the criteria for FDA oversight as a drug, device or biologic and is regulated as a Human Cells, Tissues, and Cellular and Tissue-based product (HCT/Ps) under Section 361 of the Public Health Service Act by the Food and Drug Administration (FDA). It is regulated solely under section 361 of the PHS Act and the regulation in 21 CFR 1271.10. HCT/P's regulated under section 361 PHS Act do not require an 510k, IND or BLA prior to distribution. The manufacturer of the product, Snoasis Medical LLC in Golden Colorado, properly registered the establishment and the product with the FDA (see attached screenshot) as required per 21 CFR 1271.10. The product is designed for use as wound covering in a variety of dental applications.

Quadrants (right/left, upper/lower) will randomly be assigned by block randomization via a code in an envelope with either 1) scaling and root planing alone, or 2) scaling and root planing with 8 x 8mm dHACM placement within the periodontal pocket at >5mm sites. The subject will act as his/her own control. There will be one side of the mouth that will receive the dHACM intervention with scaling and root planing and one side that will be the control (scaling and root planning only). Depending on the extent of the disease (>5mm probing depths) the intervention may involve upper and lower jaws on that side of the mouth or only one jaw per side (1-2 interventions/1-2 controls per mouth). The addition of dHACM will be a one-time placement.

The only research-related procedures that will differ from standard of care are standardizing the x-rays (with custom bite block), placement of the dehydrated human amnion-chorion membrane (dHACM), supra-gingival cleaning at 3 and 6 months (instead of supra- and sub-gingival) and x-rays taken at 9 months, 3 and 5 years. The two examiners (board certified periodontists) completing the periodontal examination will be blinded to the treatment allocated to the patient by the clinical provider (graduate periodontal resident or hygienist). Clinical measurements which are standard of care of a periodontal examination will include: probing depth, bleeding on probing, clinical attachment level, mobility, and plaque index (Sillness and Loe index). Probing measurements will be made at 6 location points on all teeth in the dentition using a calibrated University of North Carolina (UNC) periodontal probe with readings made to the nearest millimeter. Clinical attachment levels will be made from the cemento-enamel junction or nearest landmark. All sites with probing depths measuring >4mm will be measured a second time, and the average of the 2 readings will be used as the site-specific probing depth endpoint. Concomitant medications and safety evaluation will be recorded at each visit. Any suspected adverse events or allergic responses will be evaluated by the investigator.

Clinical measurements will be made at the following time points: baseline; Month 1; Month 3; Month 6; Month 9; Year 3; Year 5. Four bitewing radiographs will be taken for evaluation with custom bite mounting utilizing a long cone paralleling technique and will be made at: baseline; Month 9, Year 3, and Year 5. Baseline x-rays are the standard of care for a periodontal examination. Standardizing the x-rays with a custom bite block and re-taking the x-rays at 9 months are for research-related procedures. Subject will be instructed not to perform interproximal oral hygiene for 7 days following treatment. Following the procedure, the patients will be scheduled for periodontal maintenance at a 3-month interval. At each follow-up visit, supra-gingival plaque removal will be performed, and subjects will be instructed on the Bass brushing technique as well as the proper use of dental floss as is standard of care for oral hygiene instructions. At all end time-points of the study (9 months, 3 years, and 5 years), supra- and sub-gingival scaling will be performed as indicated for each patient. Plaque removal is the standard of care for maintaining a periodontally diseased patient. For research due to the placement of the membrane, sub-gingival cleaning will be avoided at 3 and 6 months and the cleaning will be supra-gingival only. This differs from the standard of care, which would have sub- and supra-gingival cleaning at 3 and 6 months. Cleaning will return to standard of care at 9 months, where patients will have sub- and supra-gingival cleaning.

To summarize, the standard of care will be followed for the initial x-rays, clinical measurements, scaling and root planing, and during every periodontal maintenance visits (typically at a 3-month interval). For the standard of care non-standardized x-rays are normally used. For research purposes, we will be standardizing the x-rays with a custom bite block and re-taking x-rays at all end time-points of the study (9 months, year 3, and year 5). In addition, for research purposes, we will be placing the dehydrated human amnion-chorion membrane (dHACM), and having supra-gingival cleanings at 3 and 6 months (instead of supra- and sub-gingival).

Three examiners (board certified periodontists) will be calibrated to each other for the collection of the data and interexaminer reliability will be calculated. The three examiners will be calibrated for probing depth and clinical attachment levels by reproducing clinical measurements on a single patient until the measurements are consistently within 0.5 and the percentage is 95% agreement.

Collected variables:

1. Electronic health record number
2. Demographics (age, sex, race)
3. Systemic health: subject height, weight, smoking, diabetes mellitus, and hypertension status
4. Periodontal characteristics (clinical attachment loss, probing depth, bleeding on probing, the presence of restorations)

End time-points:

• 1, 3, 6, 9 months, 3 years, 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage III and IV periodontitis (generalized moderate to severe chronic periodontitis)
* At least 4 teeth (to include at least one qualifying tooth on the right and left side of the mouth) with probing depths of 6 to 9 millimeters and bleeding on probing
* at least 18 years of age
* consent to be in the study
* non-emergent dental treatment
* American Society of Anesthesiologists (ASA) Class I or II (prticipants that are systemically healthy or have a systemic condition that is well controlled and are able to receive elective dental care)

Exclusion Criteria:

* <18 years old or >100 years old
* currently pregnant or within 6 months postpartum, nursing
* require antibiotic prophylaxis prior to dental procedures as outlined by the 2017 American Heart Association guidelines
* decisionally challenged adults
* ASA Class III or IV (patients that have non-controlled systemic conditions that are unable to have elective dental care)
* had periodontal therapy within 6 months of baseline treatment visit
* antibiotic therapy within 3 months prior to enrollment
* chronic therapy within 1 month prior to enrollment with medications that could affect periodontal status or healing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Pocket Depths | Month 9, Year 3, and Year 5
  Mean change in probing depths (using a UNC probe to measure probing depths).
Clinical Attachment Levels | Month 9, Year 3, and Year 5
  Mean change in attachment level (using a UNC probe to measure attachment levels).
Radiographic Alveolar Bone Gain | Month 9, Year 3, and Year 5
  Radiographic comparison from baseline radiograph to Month 9.

CONTACTS AND LOCATIONS:
Locations (1):
- Sangeetha Chandrasekaran, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No